CLINICAL TRIAL: NCT00436943
Title: Smoking Cessation Program: A Quality Improvement Trial in a Resident Based Outpatient Clinic
Brief Title: Smoking Cessation Program: A Quality Improvement Trial in a Resident-Based Outpatient Clinic
Status: Terminated | Type: Observational
Sponsor: Atlantic Health System (Other)
Other Study IDs: R06-12-021; Smoking Cessation
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Smoking
Keywords: smoking cessation; nicotine replacement therapy; bupropion; smoking
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy; Bupropion; Referral and Consultation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

GROUPS / COHORTS (1):
- A: Smokers
  Interventions: Drug: nicotine replacement therapy and bupropion; Behavioral: smoking cessation counseling and referrals

INTERVENTIONS:
Drug: nicotine replacement therapy and bupropion — 3-6 months
Behavioral: smoking cessation counseling and referrals — Organizational counseling and referrals

SUMMARY:
The researchers hypothesize that smoking cessation counseling improves with the implementation of a smoking status assessment data sheet in routine consults. This is a quality improvement study design to evaluate the impact of the implementation of a more formal smoking status evaluation in a resident/faculty driven outpatient clinic.

DETAILED DESCRIPTION:
We hypothesize that smoking cessation counseling improves with the implementation of a smoking status assessment data sheet in routine consults. This is a quality improvement study design to evaluate the impact of the implementation of a more formal smoking status evaluation in a resident/faculty driven outpatient clinic. This will be an observational study in which differences in quality measures will be compared between baseline and re-measurement periods. Population target: 900 patients screened before and after the implementation of the QI intervention. Primary outcome: smoking status evaluation. Secondary Outcome: number of patients advised to quit, plan implementation for smoking cessation, smoking cessation program referrals, number of NRT and bupropion prescription.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Seen at MMH family health center
* Current smoker

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2007-01; Study Completion 2008-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Harris, MD, Principal Investigator — Atlantic Health System - Morristown Memorial Hospital
Locations (1):
- Family Health Center at Morristown Memorial Hospital, Morristown, New Jersey, United States